CLINICAL TRIAL: NCT00938275
Title: Gender vs. Fed/Fasted State vs. Capsule/Liquid Suspension Formulation Study
Brief Title: A Clinical Study to Assess the Effect of Food and Gender on the Pharmacokinetics of SRT2104 Administered as an Oral Suspension or Capsule Formulation to Normal Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sirtris, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 113261
Record Dates: First submitted 2009-07-09; First posted 2009-07-13 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — SRT2104

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 0.5g SRT2104 (Experimental): Cohort 1 (10 males) & Cohort 2 (10 females) must attend the clinic on 4 separate treatment visits during the study; each treatment visit will be one week apart. At each treatment visit, subjects will receive one of the following 4 treatments:
  A) 0.5g SRT2104 administered as an oral suspension in the fasted state B) 0.5g SRT2104 administered as an oral suspension following consumption of a standard meal C) 0.5g SRT2104 administered as two 0.25g capsules in the fasted state D) 0.5g SRT2104 administered as two 0.25g capsules following consumption of a standard meal.
  For treatments A and C, subjects will have fasted for at least 10 hours overnight. Water will be restricted from 1h prior to dosing until 1h post dose. A light lunch will be provided 4h post dose. For treatments B and D, subjects will receive SRT2104 within 30 min following the start of consumption of a standardized non high-fat meal (approximately 650 kcal with approximately 30% of calories derived from fat).
  Interventions: Drug: 0.5g SRT2104

INTERVENTIONS:
Drug: 0.5g SRT2104 — SRT2104 will be supplied in two forms: as 0.5g powder which will be prepared by the pharmacist/designee into a liquid suspension and as two hard gelatin capsules, each containing 0.25g SRT2104. The dosing vehicle for the liquid suspension is 1% (by weight) hypromellose acetate succinate in water, which is used as a suspension aid and a dispersant for the SRT2104.
  Each formulation of test material will be administered orally, in a single dose to the subjects in the fasted state and following consumption of a standard meal. Neither the investigator nor the subjects enrolled will be blinded to treatment assignment.

SUMMARY:
The primary objective of this study is to assess the pharmacokinetic profile of a single 500 mg dose of SRT2104 administered as an oral suspension and a capsule formulation to normal healthy male and female volunteers in both the fed and fasted state.

The secondary objective is to assess the safety and tolerance of SRT2104 administered as an oral suspension and as a capsule formulation to healthy male and female volunteers in both the fed and fasted state.

ELIGIBILITY:
Inclusion Criteria:

* Be a healthy male or female within the age range of 18 to 55 years.
* Voluntarily sign a Research Ethics Committee (REC)-approved informed consent form to participate in the study after all relevant aspects of the study have been explained and discussed with the subject.
* Have Hematology, Coagulation, Clinical Chemistry and Urinalysis test results that are within normal, allowable limits (if out-of-range, must be considered clinically significant to be exclusionary) and performed within 21 days of receiving first dose of test material.
* Have a BMI (Body Mass Index) between 18.0 and 30.0 kg/m^2.
* Be clear of any history of HIV and hepatitis B and C.
* Have no significant disease or clinically significant abnormal laboratory value as deemed by the investigator on the laboratory evaluations, medical history, or physical exam.
* Have a normal 12-lead ECG or an ECG with abnormality considered to be clinically insignificant.
* Have the ability to communicate with the investigative site staff in a manner sufficient to carry out all protocol procedures as described.
* All subjects and their partner must agree to use an acceptable double barrier method for birth control from the Screening visit through 3 months after the last dose of test material.
* All female subjects must be of non-childbearing potential. For the purposes of this study, this is defined as the subject being amenorrheic for at least 12 consecutive months or at least 6 weeks post-surgical bilateral oophorectomy with or without hysterectomy. (Menopausal status will be confirmed by demonstrating levels of follicle stimulating hormone (FSH) of 20 - 138 mIU/ml and oestradiol < 20 pg/ml at entry. In the event a subject's menopause status has been clearly established (for example, the subject indicates she has been amenorrheic for 10 years), but FSH and/or oestradiol levels are not consistent with a post-menopausal condition, determination of subject eligibility will be at the discretion of the principal investigator following consultation with the sponsor.
* Subject agrees to refrain from consumption of grapefruits and/or grapefruit juice from 7 days prior to day -1 of treatment visit 1 through to the end of subject's final study visit.

Exclusion Criteria:

* Subject has had a major illness in the past three months or any significant ongoing chronic medical illness that the Investigator would deem unfavorable for enrollment.
* Subject has renal or liver impairment.
* Subject has a history of gastro-intestinal surgery or has a current gastrointestinal disease which may influence drug absorption.
* Subject has a history, within 3 years, of drug abuse (including Benzodiazepines, opioids, amphetamine, cocaine, and THC) or a positive drug result at Screening.
* Subject smokes more than 5 cigarettes a day.
* Subject has a history of alcoholism, and/or is currently drinking more than three drinks per day [one drink is equal to one unit of alcohol (one glass of wine, half a pint of beer, one measure of a spirit)].
* Subject has participated in a clinical trial within the past three months (defined as three months from the date of last dose of an investigational medicinal product).
* Subject has a history of difficulty in donating blood or accessibility of veins in left or right arm.
* Subject has donated blood (one unit or 350 mL) within three months prior to receiving test material.
* Subject is taking herbal products, over-the-counter medication or prescription drug therapy (with the exception of hormone replacement therapy for female subjects) for which 5 times the half-life is longer than 21 days (i.e., the Screening period) prior to enrollment into the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-01-20 (Actual); Primary Completion 2009-03-27 (Actual); Study Completion 2009-03-27 (Actual)

PRIMARY OUTCOMES:
Characterize and compare the pharmacokinetic profile of a single 500 mg dose of SRT2104 administered as an oral suspension and as a capsule formulation. | PK time points: pre-dose (0 hrs); 0.25, 0.5, 0.75, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 5.0. 6.0, 8.0, 10, 12, 15, 24, 36, 48, 72 hours post dose.

SECONDARY OUTCOMES:
Assess the safety and tolerance of SRT2104. | AEs, concomitant medications (as applicable), vital signs, physical examinations, laboratory parameters, and ECG parameters will be collected for the duration of the study.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Merthyr Tydfill, Glamorgan, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Hoffmann E, Wald J, Lavu S, Roberts J, Beaumont C, Haddad J, Elliott P, Westphal C, Jacobson E. Pharmacokinetics and tolerability of SRT2104, a first-in-class small molecule activator of SIRT1, after single and repeated oral administration in man. Br J Clin Pharmacol. 2013 Jan;75(1):186-96. doi: 10.1111/j.1365-2125.2012.04340.x. PMID 22616762
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 113261 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/113261?search=study&search_terms=113261#rs
- Available data/document: Informed Consent Form: 113261 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113261 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113261 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113261 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113261 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113261 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113261 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register